CLINICAL TRIAL: NCT02395900
Title: The Effects of Flaxseed Supplement on Lipid Profile, Liver Enzymes, Inflammatory Factors and Hepatic Fibrosis in Patients With Nonalcoholic Fatty Liver Disease
Brief Title: The Effects of Flaxseed Supplement on Biochemical Factors and Hepatic Fibrosis in Patients With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 567
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flaxseed (Active Comparator): 30 grams Flaxseed powder
  Interventions: Dietary Supplement: Flaxseed
- control (Placebo Comparator): dietary and exercise recommendation
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: Flaxseed
  Arms: Flaxseed
Other: control
  Other Names: no supplement
  Arms: control

SUMMARY:
To study the effects of Flaxseed supplement on lipid profile, liver enzymes, inflammatory factors and hepatic fibrosis in patients with Nonalcoholic Steatohepatitis (NASH), 50 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 2 and 3 will be randomly allocated to receive placebos or 30 grams Flaxseed powder for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes, some inflammatory markers, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40
* Serum alaninaminotransferase more than 1.5 fold of upper limit of normal range
* Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

* Diabetes
* Taking any kind of antibiotics two weeks before recruitment
* History of alcohol consumption
* pregnancy or lactation
* Professional athletes
* Other liver disease (viral/etc)
* Use of drugs such as calcium channel blockers, high dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs, lipid-lowering agents, metformin and vitamin E
* A history of Hypertension, Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* History of Upper GI surgery / Prior surgical procedures such as jejunoileal or jejunocolic bypass, gastroplasty
* Following program to lose weight in recent 3 mo
* A history of hypothyroidism or Cushing's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Alaninaminotransferase (ALT) | 12 weeks
Liver fibrosis | 12 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 12 weeks